CLINICAL TRIAL: NCT06111066
Title: Vitamin D Levels in Neonatal Umbilical Cord Blood: Factors and Prognostic Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-900-01
Record Dates: First submitted 2023-10-09; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Vitamin d Deficiency
Keywords: vitamin D; neonatal umbilical cord blood; influence factors; prognosis
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- vitamin D deficiency: The umbilical cord blood 25(OH)D levels: <30nmol/L
- vitamin D insufficiency: The umbilical cord blood 25(OH)D levels: 30~50nmol/L
- vitamin D sufficiency: The umbilical cord blood 25(OH)D levels: >50~250nmol/L

SUMMARY:
This study is a retrospective-prospective cohort study that investigates the factors influencing neonatal umbilical cord blood 25(OH)D levels, and the impact of exposure to low intrauterine 25(OH)D levels on neonatal prognosis. Newborns born in Sun Yat-sen Memorial Hospital of Sun Yat-sen University from August 2023 to August 2024 were selected. 2ml of umbilical cord blood was collected to test serum 25(OH)D levels. Based on the umbilical cord blood 25(OH)D levels, newborns were divided into three groups: vitamin D deficiency (<30nmol/L), insufficiency (30~50nmol/L), and sufficiency (>50~250nmol/L). Factors influencing neonatal vitamin D levels at birth were investigated by reviewing medical records, questionnaire collection, phone interviews, etc., collecting data on basic neonatal information, maternal information, complications during pregnancy, prenatal biochemical test results, medication history during pregnancy, lifestyle habits during pregnancy, and vitamin D supplementation status. Phone follow-ups on the health of the newborns during their hospital stay and at 1 month and 2 months after discharge were conducted to investigate the impact of exposure to low intrauterine 25(OH)D levels on neonatal prognosis, providing a theoretical basis for early intervention in high-risk pregnant women and early identification of high-risk groups with vitamin D deficiency or insufficiency among newborns.

Miscarriages prevention is a major feature of our hospital's obstetrics department. Many pregnant women who are hospitalized and give birth at our hospital have a history of fetus protection. Choosing pregnant women and newborns from our hospital's obstetrics department as research subjects is conducive to exploring the impact of specific diseases and medication histories on neonatal vitamin D deficiency, which is an innovative aspect of this study.

ELIGIBILITY:
Inclusion Criteria:

* Newborns delivered in Sun Yat-sen Memorial Hospital's obstetrics department.
* Relatives agree to use clinically discarded specimens for research and have signed a consent form.

Exclusion Criteria:

* Newborns with genetic mutations or congenital malformations.
* Patients who died before discharge.
* Pregnant women with conditions like chylous diarrhea, inflammatory bowel disease, and other chronic digestive system diseases.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Selected newborns and their mothers who were born at Sun Yat-sen Memorial Hospital of Sun Yat-sen University starting from September 2023.
Sampling Method: Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Maternal use of vitamin D supplements. | 2024.01-2029.12
  Investigating the situation of mothers taking vitamin D supplements during pregnancy through questionnaires and telephone interviews. This includes when they started taking them during pregnancy(weeks of gestation), the frequency of consumption(how many days a week), and the dosage taken each time(IU).
Maternal sunlight exposure. | 2024.01-2029.12
  Investigating the conditions of sunlight exposure during pregnancy through questionnaires and telephone interviews. Including ethnicity, skin color, long-term residence during pregnancy, outdoor activity time (how many hours per day), and whether sun protection measures are used when going out (such as sunscreen, umbrellas, clothing)

SECONDARY OUTCOMES:
Maternal education status. | 2024.01-2029.12
  Education levels are divided into two categories based on the highest level of education attained. The first category is 'below bachelor's degree,' which includes no formal education, elementary school, junior high school, high school, and vocational/technical education. The second category is 'bachelor's degree and above,' which includes bachelor's degrees, master's degrees, and doctoral degrees.
Maternal weight. | 2024.01-2029.12
  Calculated by maternal pre-pregnancy BMI, referring to the weight (kg) within one week before delivery, divided by the square of height (m). And the maternal weight gain during pregnancy (kg).
Pregnancy complications. | 2024.01-2029.12
  Pregnancy complications refer to health problems that occur during pregnancy. Including gestational diabetes, hypertensive disease in pregnancy, preeclampsia, intrauterine growth restriction (IUGR), and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Ouyang Ying, Prof., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No